CLINICAL TRIAL: NCT01118598
Title: To Determine if the Cardiovascular Risk Indices Including Postprandial Hypertriglyceridaemia Are Modified Favourably by Nicotinic Acid (Niacin) in Patients With Polycystic Ovary Syndrome ( PCOS)
Brief Title: Effect of Nicotinic Acid on Cardiovascular Risks Indices in Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R0920 PCOS & Niacin; ISRCTN37787683 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo arm (Placebo Comparator): this group will receive placebo as per protocol
  Interventions: Drug: placebo
- tredaptive (Active Comparator): tablet of nicotinic acid 1000 mg/laropiprant 20 mg one tablet of for 4 weeks followed by two tablets od for 8 weeks
  Interventions: Drug: tredaptive (nicotinic acid/ laropiprant)

INTERVENTIONS:
Drug: tredaptive (nicotinic acid/ laropiprant) — tablet of nicotinic acid 1000 mg/laropiprant 20 mg one tablet of for 4 weeks followed by two tablets od for 8 weeks
  Other Names: tredaptive
  Arms: tredaptive
Drug: placebo — placebo tablet one a day for first 4 weeks followed by two a day for 8 weeks
  Arms: placebo arm

SUMMARY:
Niacin will improve postprandial hyperlipidaemia and cardiovascular risks indices via its lipid lowering as well as via pleiotropic effects in patients with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a common hormone problem in young women and, as a result of it, they can experience irregular periods, reduced fertility, acne and increased body hair. Frequently, increased weight is a feature. Research suggests that they could have a higher risk of diabetes, high cholesterol and cardiovascular disease such as high blood pressure, angina, heart attack and stroke.

The fat from the diet is transported from the stomach into the blood and then taken up by the liver, muscles and fat tissues to store or use as an energy source. Delayed removal of fat from the circulation resulting rise of fat after a meal has been known to happen in PCOS. High fats after a meal are a strong risk factor for cardiovascular disease.

Niacin has been in clinical use to lower bad cholesterol and to increase good cholesterol for many years. It has been proved to be effective in reducing risks of heart disease in patients with diabetes. However the effect of niacin on reducing cardiovascular risks and reducing fat level after a meal in PCOS has not been studied and this is why we plan to do this research.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 - 50 years
* Has polycystic ovary syndrome diagnosed according to Rotterdam consensus statement

Exclusion Criteria:

* Pregnancy/trying to conceive/breast feeding
* History of cardiovascular, renal, hepatic and active thyroid disease
* History of gout
* History of alcohol abuse
* History of diabetes
* History of allergy to nicotinic acid/laropiprant or food
* History of bleeding disorders/active peptic ulcers
* Patient on antihypertensive medications
* Patient on anticoagulants
* Patient on any hormonal replacement or oral contraceptive pills or cholesterol lowering agents
* History of smoking more than 15 pack year
* Unwilling for GP to be informed

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Reduction in postprandial triglyceride | 3 months
  Postprandial triglyceride will be measured using meal test.

SECONDARY OUTCOMES:
Reduction in high sensitivity C-reactive protein (CRP) | 3 months
Improvement in peripheral arterial tone (PAT- index) | 3 months
  Peripheral arterial tone (PAT- index) will be measured using ENDO PAT 2000 before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Atkin, FRCP, PhD, Principal Investigator — University of Hull
Locations (1):
- Hull & East Yorkshire Hospitals NHS Trust, Hull, United Kingdom

REFERENCES:
- [Result] Aye MM, Kilpatrick ES, Afolabi P, Wootton SA, Rigby AS, Coady AM, Sandeman DD, Atkin SL. Postprandial effects of long-term niacin/laropiprant use on glucose and lipid metabolism and on cardiovascular risk in patients with polycystic ovary syndrome. Diabetes Obes Metab. 2014 Jun;16(6):545-52. doi: 10.1111/dom.12255. Epub 2014 Feb 9. PMID 24401089